CLINICAL TRIAL: NCT06737666
Title: Effects of Tong-Xie-Yao-Fang in Regulating Treg/Th17 Imbalance of Diarrhea-predominant Irritable Bowel Syndrome by Trp-Kyn-AhR Pathway
Brief Title: Study on the Effectiveness and Mechanism of Tong-Xie-Yao-Fang in Treating Diarrhea-predominant Irritable Bowel Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022XLA162-3
Record Dates: First submitted 2024-09-28; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tong-Xie-Yao-Fang intervention group (Experimental)
  Interventions: Drug: Tong-Xie-Yao-Fang
- healthy people (No Intervention)

INTERVENTIONS:
Drug: Tong-Xie-Yao-Fang — Tong-Xie-Yao-Fang granules were taken 2 bags at a time, 2 times per day at 1h after meal for 4 weeks.
  Arms: Tong-Xie-Yao-Fang intervention group

SUMMARY:
Traditional Chinese Medicine focuses on the main pathogenesis of liver depression and spleen deficiency, and treats them from the perspective of soothing the liver and strengthening the spleen to treat on Diarrhea-predominant irritable bowel syndrome (IBS-D) . The classic formula for treating is the Tong-Xie-Yao-Fang (TXYF). Based on metabolomics and metagenomics, the research group studied the intestinal flora and host co metabolism of TXYF in the treatment of diarrhea predominant IBS-D, in order to clarify the mechanism of TXYF in the treatment of IBS-D.

DETAILED DESCRIPTION:
Diarrhea-predominant irritable bowel syndrome (IBS-D) is a common clinical functional gastrointestinal disease with unclear mechanism, which is mostly induced by emotion. There is no specific treatment for this disease. Traditional Chinese Medicine focuses on the main pathogenesis of liver depression and spleen deficiency, and treats them from the perspective of soothing the liver and strengthening the spleen. The classic formula for treating is the Tong-Xie-Yao-Fang (TXYF).Previous studies of our research group have shown that TXYF can significantly improve the symptoms of abdominal pain and diarrhea in patients with IBS-D, and improve the quality of life of patients. The effectiveness and safety of TXYF in the treatment of IBS-D have been evaluated, and its mechanism of action has also been explored.Modern studies have shown that changes in the local immune microenvironment can affect intestinal immunity and neuroregulation, mucosal barrier damage and abnormal co-metabolism of flora and host, which may be important reasons for the occurrence and development of IBS-D, but the detailed mechanism is unclear.Therefore, based on metabolomics and metagenomics, the research group studied the intestinal flora and host co metabolism of TXYF in the treatment of diarrhea predominant IBS-D, in order to clarify the mechanism of TXYF in the treatment of IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* IBS-D patients and healthy volunteers meeting diagnostic criteria;
* Aged between 18 and 70;
* Have not taken antibiotics, steroids and other hormones, Chinese herbal preparations (including oral and intravenous injections), microecological preparations or probiotics such as yogurt in the past week.
* Patients sign informed consent forms and are willing to receive appropriate treatment, and volunteers are willing to cooperate in taking blood, urine, stool and other samples.

Exclusion Criteria:

* Patients with serious heart, liver, kidney and other major organ diseases, hematopoietic system, nervous system or mental diseases;
* Other organic diseases of the digestive system (such as peptic ulcers), organic diseases such as tumors indicated by recent colonoscopy, or systemic diseases affecting digestive motility (such as hyperthyroidism, diabetes);
* Need to continue to use drugs that may affect gastrointestinal function (antidiarrheals, antidepressants, anti-anxiety drugs, intestinal flora regulation drugs, antibiotics, etc.);
* Have a history of drug allergy or severe food allergy for research purposes;
* Patients under 18 years of age or over 75 years of age and pregnant or lactating women;
* Severe negative life events occurred during treatment;
* There is currently any form of psychotherapy in progress;
* No intention to cooperate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fecal metagenomic detection of bacteria associated with Trp metabolism | 16weeks
Serum detection by Elisa | 16weeks
Serum Trp metabolism was measured by metabolomics | 16weeks
Th17/Treg ratio in peripheral blood was measured by flow cytometry | 16weeks
Colon tissue was detected by immunofluorescence and histochemistry analysis | 16weeks
  Foxp3 ,RORrt ,AhR ,IDO1 ,Tyn

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China